CLINICAL TRIAL: NCT06515574
Title: Effect of Developmental Care on Very Low Birth Weight Infants: a Stepped-wedge Cluster Randomised Trial
Brief Title: Effect of Developmental Care on Very Low Birth Weight Infants
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Supportive Care
Other Study IDs: 20240610
Record Dates: First submitted 2024-07-10; First posted 2024-07-23 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Intervention
Keywords: developmental care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Developmental care (Experimental): In stage 1, participant in this arm will receive the developmental care
  Interventions: Behavioral: developmental care
- Usual care (No Intervention): Participant in this arm will receive the usual care

INTERVENTIONS:
Behavioral: developmental care — Individualized Developmental Care that includes the light, noise, sleep, etc.
  Arms: Developmental care

SUMMARY:
The goal of this clinical trial is to learn if developmental care works when implemented in very low birth weight infants. The main questions it aims to answer are:

* Does developmental care shorten the length of hospital stay in the very low birth weight infants?
* Does developmental care increase the opportunity of family centered care in the very low birth weight infants? The clinical trial will use a 36-month stepped-wedge cluster-randomised trial conducted across 40 Neonatal intensive care units . A developmental care bundle will be tailored to meet the identified needs of participating NICUs.

DETAILED DESCRIPTION:
Developmental care in the NICU focuses on creating a nurturing environment that supports the physical, emotional, and developmental needs of premature infants. This approach includes strategies like minimizing unnecessary noise and light, ensuring appropriate positioning and handling of infants, promoting skin-to-skin contact, and facilitating parental involvement in care.

The clinical trial investigates the effectiveness of developmental care in very low birth weight (VLBW) infants. The primary objectives are to determine whether developmental care can (1) reduce the length of hospital stay and (2) enhance the opportunity for family-centered care in these infants. The study employs a 36-month stepped-wedge cluster-randomised trial design, involving 40 Neonatal Intensive Care Units (NICUs).

In this trial, all NICUs will eventually receive the intervention, but the order in which they start implementing the developmental care bundle will be randomized. This approach allows each NICU to serve as its own control, comparing outcomes before and after the intervention.

Data collection will occur at multiple time points before and after the implementation of the developmental care bundle, enabling a comprehensive analysis of its impact. By tailoring interventions to each NICU's specific context and needs, the study aims to generate robust evidence on the benefits of developmental care for VLBW infants and their families.

ELIGIBILITY:
Inclusion Criteria

1. Birth weights less than 1500 g
2. Admitted or transported to a level III NICU within 24h of birth
3. OI>30

Exclusion Criteria:

1. Severe congenital malformations
2. various chromosomal disorders
3. genetic metabolic diseases,
4. severe neurological disorders

Ages: 0 Days to 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1600 (Estimated)
Dates: Start 2024-08-30 (Actual); Primary Completion 2027-08-30 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Length of hospital stay | From the day admitted into the NICU until day on discharge, generally assessed up to 1 year
  Length of hospital stay (in days)

SECONDARY OUTCOMES:
Skin to skin care duration | From the day admitted into the NICU until day on discharge, generally assessed up to 1 year
  Skin-to-skin care, also known as kangaroo care, involves placing a newborn baby directly on a parent's bare chest. Record the duration of skin to skin care every day during the hospitalization by hours

OTHER OUTCOMES:
Parental involvement duration | From the day admitted into the NICU until day on discharge, generally assessed up to 1 year
  Parental involvement in our study is defined as the parents take part in the daily Care Activities (diapering, bathing, clothing and feeding for their babies).Record the duration of parental involvement every day during the hospitalization by hours

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Children's hospital of Fudan university, Shanghai, Shanghai / 上海
  - Children's Hospital of Fudan University, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: Yes
Unidentified individual participant data (including data dictionaries) will be made available, in addition to study protocols, the statistical analysis plan, the informed consent form and the related code. The data will be made available upon publication to researchers who provide a methodologically sound proposal for use in achieving the goals of the approved proposal. Proposals should be submitted to corresponding authors.